CLINICAL TRIAL: NCT05341297
Title: Digital Parent-led Transdiagnostic Interventions for Child and Adolescent Anxiety and Depressive Disorders
Brief Title: A Transdiagnostic Internet Intervention for Parents of Children With Anxiety and Depressive Symptoms
Acronym: ParentKIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Costina-Ruxandra Păsărelu, Assistant professor, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GTC 31371/2020
Record Dates: First submitted 2022-04-11; First posted 2022-04-22 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Emotional Problem; Anxiety; Depression; Psychological Distress
Keywords: Internet intervention; transdiagnostic; parent-led intervention; internalizing problems; children; Rational emotive and behavioral therapy
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ParentKIT (Experimental): Transdiagnostic parent-led Internet-delivered intervention Participants in the experimental group will have access to the ParentKIT intervention. The intervention was developed based on existing Cognitive Behavioral Therapy/ Rational Emotive Behavior Therapy protocols for parents of children with internalizing problems. It consists of nine modules delivered over three weeks.
  Interventions: Behavioral: ParentKIT
- Waitlist (No Intervention): Participants in the waitlist condition will have access to the program after 3 weeks.

INTERVENTIONS:
Behavioral: ParentKIT — The intervention is structured in 9 modules through which parents learn to identify and manage their children's anxiety and depressive symptoms. The Internet intervention is guided by two psychotherapists under supervision training in Cognitive Behavioral Therapy, trained by the first author on the treatment protocol.
  Arms: ParentKIT

SUMMARY:
The purpose of this study is to evaluate the efficacy of a transdiagnostic, parent-led, Internet-delivered intervention in reducing child and adolescent internalizing problems.

DETAILED DESCRIPTION:
Anxiety and depressive symptoms are common in children and adolescents. There is substantial research indicating that transdiagnostic Internet interventions are effective for adults and children with anxiety and depressive disorders; however, there is limited research on the efficacy of such programs aimed at parents of children and adolescents with anxiety and depressive symptoms. This study aims to investigate the efficacy of a transdiagnostic Internet intervention for parents of children with elevated anxiety and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* parent of a child/ adolescent aged 6 to 14 years
* elevated internalizing problems
* have Internet access

Exclusion Criteria:

* undergoing psychotherapy/ pharmacological treatment

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the brief Revised Children's Anxiety and Depression Scale - parent version | Baseline, 3 weeks and follow-up at 1 month after treatment termination
  Measure of child anxiety and depressive symptoms, as reported by parents. Scores range between 0 and 33; higher scores indicate higher anxiety and depressive symptoms.

SECONDARY OUTCOMES:
Change in the Patient Health Questionnaire-4 | Baseline, 3 weeks and follow-up at 1 month after treatment termination
  Measure of anxiety and depressive symptoms - will be used to measure changes in parental distress. Scores range between 0 and 12. Higher scores indicate higher distress.
Change in the Parental Self-Efficacy Scale | Baseline, 3 weeks and follow-up at 1 month after treatment termination
  Measure of parental self-efficacy in relationship to parenting practices that may decrease anxiety and depression risks for adolescents. Total scores range between and 9 and 36. Higher scores indicate higher parental self-efficacy.
Change in the Family Accommodation Scale | Baseline, 3 weeks and follow-up at 1 month after treatment termination
  Measure of parental anxiety accommodations. Scores range between 0 and 52. Higher scores indicate higher parental anxiety accommodations.
Satisfaction with the intervention | 3 weeks after treatment initiation
  Client satisfaction will be measured with Client Satisfaction Questionnaire, short form (Attkisson & Zwick, 1982). Scores range from 8 to 32, with higher scores indicating greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Costina R Păsărelu, Ph.D, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be uploaded after publication of the results.
Time Frame: De-identified data will be uploaded after publication of the results.
Access Criteria: Upon the completion of the study, de-identified datasets will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Poetar CR, Dobrean A, Andersson G. Preliminary efficacy of a transdiagnostic parent-led internet-delivered intervention for children with anxiety and depressive symptoms: a pilot randomized controlled trial. Child Adolesc Psychiatry Ment Health. 2024 Mar 6;18(1):31. doi: 10.1186/s13034-024-00721-3. PMID 38448874